CLINICAL TRIAL: NCT02643628
Title: A Pilot Study to Evaluate the Safety and Effectiveness of Microneedling and Bellafill to Treat Facial Acne Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suneva Medical, Inc. (Industry)
Collaborators: ethica Clinical Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUN-1503
Record Dates: First submitted 2015-12-29; First posted 2015-12-31 (Estimated); Results first posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-09

CONDITIONS: Atrophic Acne Scars
MeSH Terms: interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Microneedling Only (Experimental): All eligible scars within the treatment areas on each side of the face will receive microneedling treatment. The device will be rolled in a horizontal direction with medium pressure. After every roll, the device will be lifted and positioned a few millimeters inferior to the previous starting point. Rolling will be repeated until the entire skin area has been treated. The device will then be reoriented vertically and rolling will be repeated in a vertical direction.
  Interventions: Procedure: Microneedling
- Microneedling followed by Bellafill treatment (Experimental): Subjects undergo microneedling as described for the Microneedling Only group. Then at Week 12, all eligible scars within the treatment areas on each side of the face will be treated with Bellafill (injected using a standard tunneling technique). A touch-up treatment is allowed at Month 1 after initial treatment, if additional treatment is required to achieve optimal correction.
  Interventions: Device: Microneedling followed by Bellafill treatment

INTERVENTIONS:
Procedure: Microneedling
  Arms: Microneedling Only
Device: Microneedling followed by Bellafill treatment
  Arms: Microneedling followed by Bellafill treatment

SUMMARY:
This is an open-label, randomized, multicenter, prospective trial assessing the efficacy and safety of microneedling treatment alone vs. microneedling treatment followed by treatment with Bellafill for correction of distensible atrophic facial acne scars.

DETAILED DESCRIPTION:
The study is divided into two study Periods. In Period I, subjects will attend a Screening visit (Week -4) and undergo the Bellafill skin test. At Visit 1 (Day 0), all subjects will commence microneedling treatment for their atrophic acne scars. Subjects will then return to the clinic at Week 3 and Week 6 (Visits 2 and 3, respectively) for follow-up evaluation and additional cycles of microneedling treatment.

At Week 12 (Visit 4), all subjects commence Period II and are randomized to Bellafill Treatment (Track A) or to No Treatment (Track B):

* Track A: Consists of three (3) study visits. At Visit 4, subjects randomized to the "Bellafill" group will receive treatment with Bellafill for their atrophic acne scars. Subjects return for Visit 5A (Month 1 after randomization) for evaluation and follow-up, and will receive touch-up injections with Bellafill to achieve optimal correction (if necessary). Subjects will then be followed-up at Visits 6A and 7A which will occur at Month 3 and Month 6, respectively, after their last Bellafill treatment.
* Track B: Consists of one (1) study visit. At Visit 4, subjects randomized to the "No Treatment" group will complete visit evaluations and then return for follow-up at Visit 5B (approx. Month 3 after randomization).

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, male or female subjects of any race, 21 years of age or older. Female subjects of childbearing potential must have a negative urine pregnancy test result at Baseline and practice a reliable method of contraception throughout the study.
* Negative response to the Bellafill Skin Test.
* Presence of ≥4 distensible atrophic acne scars located within the facial treatment area. Subject desires correction of his/her atrophic acne scarring.
* All Fitzpatrick skin types are eligible.
* Subjects with a history of HSV-1 (oral herpetic outbreak) willing to accept prophylactic treatment with antiviral medication.
* Willing to withhold additional aesthetic therapies to the proposed treatment area (e.g., other soft tissue fillers such as hyaluronic acid, and/or any resurfacing procedures (as described in Protocol Section 5.3) for the duration of the study.
* Able to follow study instructions and likely to complete all required visits, as assessed by the Investigator.
* Sign an IRB-approved Informed Consent Form, Photographic Release Form, and the Authorization for Use and release of Health and Research Study Information (HIPAA) Form prior to any study-related procedures being performed.

Exclusion Criteria:

* Female subjects that are pregnant (positive urine pregnancy test), breast-feeding, or who are of childbearing potential and not practicing a reliable method of birth control.
* Undergone facial treatments with any prohibited treatment/procedures and/or use of any other prohibited treatment/procedure.
* Excisional facial surgery (such as Blepharoplasty, Face Lift, Rhinoplasty) of the face ≤ 6 months prior to study enrollment or plans for facial surgery during the study.
* History of bleeding disorders.
* Presence of any skin pathology or condition that could interfere with the evaluation of the treatment areas, worsen due to the proposed treatment or require interfering topical, systemic or surgical therapy.
* Recent or current history of inflammatory skin disease, infection, cancerous/pre-cancerous lesion, unhealed wound or clinically significant acne in the proposed treatment areas. Clinically significant acne is defined as a patient whom has ≥3 active inflammatory acne lesions in the treatment areas.
* History of systemic granulomatous diseases active or inactive (e.g., Sarcoid, Wegeners, TB) or connective tissue diseases (e.g., lupus, dermatomyositis).
* Hypertrophic acne scars, any evidence of keloid scarring in the treatment area.
* Known hypersensitivity or previous allergic reaction to any of the components of the study device (including lidocaine or any amide-based anesthetic), or has a history of allergies to any bovine collagen products, including but not limited to injectable collagen, collagen implants, hemostatic sponges, and collagen-based sutures.
* Undergone or be planning to undergo desensitization injections to meat products.
* Unable to communicate or cooperate with the Investigator due to a language barrier (non-English speaking), poor mental development, or impaired cerebral function.
* Evidence of alcohol or drug abuse (Investigator opinion), or history of poor cooperation, non-compliance with medical treatment, or unreliability.
* Use of an investigational device, biologic or drug in the past 30 days, or be currently participating in an experimental drug, biologic or device trial.
* Exhibits additional physical attributes which prevent the assessment or treatment of the atrophic scars, as judged by the Investigator, such as excessive hair, traumatic or surgical scars, excessive hyperpigmentation in the treatment area, etc.
* Has a condition or be in a situation that, in the Investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.
* An employee (or a relative of an employee) of the Investigator, Sponsor or representative of the Sponsor.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-10-10 (Actual); Primary Completion 2017-06-05 (Actual); Study Completion 2017-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Seretta, Study Director — Suneva Medical
Locations (1):
- Call Suneva for Info, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 55 subjects screened with 45 meeting eligibility criteria and enrolled. One subject discontinued by investigator. 44 subjects randomized 23 to Microneedling + Bellafill and 21 to Microneedling alone.
Groups:
- Microneedling Only: All subjects eligible scars within the treatment areas on each side of the face will receive microneedling treatment. At Week 12 subjects randomized to no further treatment.
- Microneedling Followed by Bellafill Treatment: All Subjects undergo microneedling as described for the Microneedling Only group. Then at Week 12, all eligible scars within the treatment areas on each side of the face will be treated with Bellafill (injected using a standard tunneling technique). A touch-up treatment is allowed at Month 1 after initial treatment, if additional treatment is required to achieve optimal correction.
  Microneedling followed by Bellafill treatment
Period: Overall Study
Arm/Group | Microneedling Only | Microneedling Followed by Bellafill Treatment
Started | 21 | 23
Completed | 20 | 17
Not Completed | 1 | 6
Not completed — Lost to Follow-up | 1 | 4
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Relocated out of state | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Microneedling Only: All eligible scars within the treatment areas on each side of the face will receive microneedling treatment. Subjects randomized at week 12 to no further treatment.
- Microneedling Followed by Bellafill Treatment: Subjects undergo microneedling as described for the Microneedling Only group. Then at Week 12, all eligible scars within the treatment areas on each side of the face will be treated with Bellafill (injected using a standard tunneling technique). A touch-up treatment is allowed at Month 1 after initial treatment, if additional treatment is required to achieve optimal correction.
  Microneedling followed by Bellafill treatment
- Total: Total of all reporting groups
Arm/Group | Microneedling Only | Microneedling Followed by Bellafill Treatment | Total
Number analyzed (Participants) | 21 | 23 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 23 | 44
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.50 (10.68) | 40.67 (13.12) | 38.68 (12.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 18 | 29
  Male | 10 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 10
  Not Hispanic or Latino | 14 | 20 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 1 | 1 | 2
  White | 17 | 17 | 34
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 23 | 44

OUTCOME MEASURES:

1. Primary Outcome: Acne Scar Assessment Scale (ASAS)
Description: • Acne Scar Assessment Scale (ASAS): a validated 5-point static scale assessing physician impression of acne scar severity where as 1=clear and 5 = severe
Time Frame: 6 months post-injection for Bellafill arm. 3 months Microneedling alone arm
Population: All subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Microneedling Only: All eligible scars within the treatment areas on each side of the face will receive microneedling treatment. The device will be rolled in a horizontal direction with medium pressure. After every roll, the device will be lifted and positioned a few millimeters inferior to the previous starting point. Rolling will be repeated until the entire skin area has been treated. The device will then be reoriented vertically and rolling will be repeated in a vertical direction.
  Microneedling
Arm/Group | Microneedling Followed by Bellafill Treatment | Microneedling Only
Number analyzed (Participants) | 17 | 19
units on a scale | 2.65 (0.75) | 3.71 (0.75)

2. Primary Outcome: Physician Global Aesthetic Improvement Scale (PGAIS)
Description: The PGAIS is used for the physician to rate the improvement of the acne scar. 5 point Likert Scale ranging from 5 to 1 with 5 = Much Improved and 1 = Much Worse
Time Frame: From week 12 to 6-months for the Treatment arm and 3 months for the Microneedling only arm
Population: There were 21 subjects in the microneedling arm however data only available for 19 subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Microneedling Only | Microneedling Followed by Bellafill Treatment
Number analyzed (Participants) | 19 | 17
units on a scale | 0.05 (0.62) | 0.35 (0.49)

3. Primary Outcome: Subject Global Aesthetic Improvement Scale (SGAIS)
Description: The SGAIS is used for the subject to rate the improvement of the acne scar. 5 point Likert Scale ranging from 5 to 1 with 5 = Much Improved and 1 = Much Worse
Time Frame: From week 12 to 6-months for the Treatment arm and 3 months for the Microneedling only arm
Population: There were 21 subjects in the microneedling arm however data only available for 19 subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Microneedling Only | Microneedling Followed by Bellafill Treatment
Number analyzed (Participants) | 19 | 17
units on a scale | 0.05 (0.62) | 0.18 (0.39)

4. Primary Outcome: Quality of Life Impact Scar (QOLIS)
Description: Quality of Life Scar Impact Scale questionnaire was used to allow the subject to specifically address how acne scarring has affected his/her emotional and functional status. Subjects completed 33 questions ratings between 1 and 7 one being less severe 4 neutral and 7 more severe. Scores are averaged for a total range of 1-7.
Time Frame: 6-months for the Treatment arm and 3 months for the Microneedling only arm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Microneedling Only | Microneedling Followed by Bellafill Treatment
Number analyzed (Participants) | 20 | 17
units on a scale | 3.90 (1.45) | 2.47 (1.42)

5. Primary Outcome: Number of Subjects With Adverse Events
Time Frame: 6-months
Measure: Count of Participants; unit: Participants
Arm/Group | Microneedling Followed by Bellafill Treatment | Microneedling Only
Number analyzed (Participants) | 23 | 21
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: six (6) months
Arm/Group | Microneedling Followed by Bellafill Treatment | Microneedling Only
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/21
Other Adverse Events (participants affected / at risk) | 2/23 | 1/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Microneedling Followed by Bellafill Treatment (N=23) | Microneedling Only (N=21)
Treatment Site Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Treatment Site Dermatitis was attributed to the microneedling procedure.
Peripheral edema of the foot (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
slight cold (Immune system disorders) | 1 (1) | 0 (0) — Subject had a slight cold

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-11): https://cdn.clinicaltrials.gov/large-docs/28/NCT02643628/Prot_SAP_000.pdf